CLINICAL TRIAL: NCT01181791
Title: Pilot Study to Evaluate the Effects of Lactobacillus Reuteri in Preterm Newborns
Brief Title: Effects of Lactobacillus Reuteri in Premature Infants
Acronym: Reuteri
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University of Miami (Other)
Collaborators: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Teresa del Moral, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20090924
Record Dates: First submitted 2010-08-02; First posted 2010-08-13 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Premature Infant Disease
Keywords: probiotics; premature infants; feeding tolerance
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Administration of probiotic Lactobacillus Reuteri
Who Masked: Participant, Care Provider, Investigator
Masking Description: Administration of placebo
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotic group (Experimental): Lactobacillus reuteri will be given at a dose of 1x108 colony forming units (CFU)/day
  Interventions: Dietary Supplement: Lactobacillus reuteri
- Placebo (Placebo Comparator): The placebo consists of an identical formulation except that the L. reuteri is not present.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — Lactobacillus reuteri DSM will be given at a dose of 1x108 colony forming units (CFU)/day
  Arms: probiotic group
Other: Placebo — The placebo consists of an identical formulation except that the L. reuteri is not present.
  Arms: Placebo

SUMMARY:
This application a phase II clinical trial to address the possible active mechanisms of probiotics and to obtain preliminary efficacy and safety data after the administration of a probiotic, Lactobacillus reuteri a population of premature infants.

The hypothesis is that the exogenous supplementation Lactobacillus reuteri to premature infants will lead to clinical beneficial effects by modifying their intestinal microbiota and enhancing their intestinal immunological response.

DETAILED DESCRIPTION:
The primary outcome "days to achieve full feeds" will be measure during the the first month of life Secondary outcomes will be measured at baseline (before intervention), 3 weeks after intervention, once intervention discontinued and at 6 months of live

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns admitted to the neonatal intensive care units with a birth weight 700-1500 g and who survive more than 3 days

Exclusion Criteria:

* Chromosomal anomalies.
* Major congenital anomalies (complex cardiac anomalies, congenital hydrocephalus, renal dysplasia)
* Congenital (e.g. jejunal atresia) and acquired (e.g. GI perforation) gastrointestinal pathology precluding oral feed and/or requiring major surgical or medical intervention
* Parental refusal
* Prior enrollment into a conflicting clinical trial

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2010-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Time to reach full feeds | First 40 days after birth
  Days to reach full feeds from the day feeds are started

SECONDARY OUTCOMES:
Intestinal colonization | 0-6 months after birth
  PCR quantification of lactobacillus reuteri in the stools
Intestinal immunological response | 0-6 months
  Quantification immunological markers in the stools

CONTACTS AND LOCATIONS:
Overall Officials: Teresa del Moral, MD, MPH, Principal Investigator — University of Miami
Locations (2):
- Chile (2):
  - Hospital Sotero del Rio, Santiago
  - Pontifica Universidad Catolica, Santiago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharif S, Meader N, Oddie SJ, Rojas-Reyes MX, McGuire W. Probiotics to prevent necrotising enterocolitis in very preterm or very low birth weight infants. Cochrane Database Syst Rev. 2023 Jul 26;7(7):CD005496. doi: 10.1002/14651858.CD005496.pub6. PMID 37493095
- [Derived] Sharif S, Meader N, Oddie SJ, Rojas-Reyes MX, McGuire W. Probiotics to prevent necrotising enterocolitis in very preterm or very low birth weight infants. Cochrane Database Syst Rev. 2020 Oct 15;10(10):CD005496. doi: 10.1002/14651858.CD005496.pub5. PMID 33058137